CLINICAL TRIAL: NCT03053739
Title: Randomized Controlled Trial to Compare the Efficacy of Combination Therapy vs Monotherapy for Pulmonary Arterial Hypertension in Systemic Sclerosis
Brief Title: To Compare the Efficacy of Combination Therapy vs Monotherapy for Pulmonary Arterial Hypertension in Systemic Sclerosis
Acronym: BosSilSS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, DR PREKSHA DWIVEDI, SENIOR RESIDENT,CLINICAL IMMUNOLOGY AND RHEUMATOLOGY ,DEPT OF INTERNAL MEDICINE, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MK/2927/DM/9430
Record Dates: First submitted 2016-12-29; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Associated Pulmonary Arterial Hypertension
Keywords: Systemic sclerosis, Associated Pulmonary Arterial Hypertension
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Sildenafil Citrate; Bosentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination arm A-Sildenafil and Bosentan (Active Comparator): Combination Arm A -Intervention- Drug
  * Tab Sildenafil 20 mg - three times a day for 6 months,and
  * Tab Bosentan 62.5mg - twice a day for 6 months
  Interventions: Drug: Sildenafil 20mg and Bosentan 62.5mg
- Monotherapy arm-Sildenafil and Placebo (Placebo Comparator): Monotherapy arm B Intervention-Drugs Tab Sildenafil 20mg- three times a day for 6 months, and Placebo tab (matched for bosentan) for 6 months
  Interventions: Drug: Sildenafil 20mg and Placebo

INTERVENTIONS:
Drug: Sildenafil 20mg and Bosentan 62.5mg — Sildenafil 20 mg three times a day and bosentan 62.5mg two times a day
  Arms: Combination arm A-Sildenafil and Bosentan
Drug: Sildenafil 20mg and Placebo — Sildenafil 20 mg three times a day and placebo (matched for bosentan)two times a day
  Arms: Monotherapy arm-Sildenafil and Placebo

SUMMARY:
The study will be carried out on 50 consecutive consenting patients of systemic sclerosis with PAH recruited from outpatient department of internal medicine and rheumatology clinic of PGIMER, Chandigarh, India It is a single centre double blind randomised controlled trial evaluating the effect of upfront dual therapy (sildenafil and bosentan) vs monotherapy (sildenafil) Participants will be randomised in 1:1 ratio to one of treatment arms. Placebo and PDE-5 inhibitors 20 mg BD to 60 mg if patient tolerates the drug well to one study arm and PDE-5 inhibitors plus ER antagonist 62.5 to max of 125 to other study group

DETAILED DESCRIPTION:
All patients fulfilling the SSc classification criteria of American College of Rheumatology during the study period will be screened for presence of PAH. Diagnosed cases of PAH based on CD echo with PAP >35mmHg based on echocardiography will be enrolled in study.Baseline NYHA functional class and 6 min walk distance in meters will be assessed. Heamogram and LFT will be measured Patients will be assessed at two weeks for side effects/safety issues. 6MWT and NYHA functional class will be reassessed at 3 months and 6 months.2D echo will be done at 6 months to measure mPAP RandomizationAll eligible patients will be randomized in a 1:1 ratio in blocks of ten between the two arms. Randomization will be stratified based on severity of PAH. The drugs will be labelled as A and B randomly by another staff member, who will not be involved in deciding the treatment of the study subjects. The randomization sequence will be generated using computer random number generator.

Blinding will be ensured by matching placebo for ERA in one group and will labelled one treatment arm as 'A' and other treatment arm as 'B'. Allocation concealment will be ensured by means of enclosing the randomization sequence in sealed opaque envelopes. Sealed opaque envelopes will contain Code 'A' or Code 'B'.

Intervention-The study consists of two treatment arms. The study drugs mainly Bosentan and Placebo will be packed into matching tablets at the dosage 62.5 mg. One treatment arm will contain Sildenafil and Placebo while other treatment arm will contain Sildenafil and Bosentan. Treatment will be initiated as 20 mg twice a day for Sildena-fil in combination with placebo once a day in one treatment arm and with Bosentan 62.5 mg once a day in other treatment arm .Dose of Sildenafil will be increased to 20 mg thrice a day at four weeks and that of Bosentan to 62.5 mg twice a day. Placebo will be also be provided twice a day.This will be continued till end of study period.. Dose adjustments in case of adverse events will be made depending on the severity of adverse events.

Statistical analysis- Intention to treat analysis will be carried for the primary and secondary outcomes. For continuous outcomes, unpaired t-test and for dichotomous outcomes chi-squares test with Yate's correction will be used. P<0.05 will be considered significant

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years
* Patients with systemic sclerosis
* PAH diagnosed as PAP>35mmHg
* NYHA functional class II,III,IV
* SSc disease duration >1years

Exclusion Criteria:

* Forced vital capacity <60% predicted
* Renal insufficiency
* Left heart disease and other relevant cardiac conditions
* Pregnant or breastfeeding female
* Patients on PAH specific therapy
* Liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pulmonary artery pressures | Baseline and 6 months
  Change in Pulmonary artery pressures measured by echocardiography at baseline and 6 months in patients of systemic sclerosis with PAH when treatment with Single(PDE-5inhibitors at dose of 20 mg maximum upto 60mg) versus Dual therapy(PDE-5inhibitors and ER antagonist 62.5 mg maximum upto 125mg) for 6 months

SECONDARY OUTCOMES:
1.Change in 6 Minute walk distance | Baseline and 6 months
  1. To compare change in 6 MWD at baseline, and 6 months when treated with single versus dual therapy.
Time To Clinical Worsening (TTCW) | Baseline and 6 months
  To compare time to clinical worsening (TTCW) in SSc patients when treated with single versus dual therapy. TTCW is defined as first occurrence of all cause deaths, PAH related hospitalisation, worsening of symptoms defined as a decrease of >15% in 6 min walk distance and worsening of NYHA functional class.
Emergent side effects of Sildenafil and Bosentan | Baseline to 6 months
  To compare the emergent side effects of sildenafil and bosentan by way of comparison of serious and nonserious side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Nandita Kakker, M.D, Study Chair — Institutional ethics committee,PGIMER Chandigarh,India
Locations (1):
- Dr Preksha Dwivedi, Chandigarh, India